CLINICAL TRIAL: NCT06688968
Title: Observational Pilot Study of Neuropsychological Profiles and Musical Engagement in Parkinson's and Alzheimer's Disease. What Are the Effects of Mnestic or Hedonic Impairment on Emotion, Reminiscence and Musical Enjoyment
Brief Title: Neuropsychological Profiles and Musical Engagement in Parkinson's and Alzheimer's Disease
Acronym: MUSENGAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Laboratoire EPSYLON (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL23_0427
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease, Early Onset; Parkinsons Disease with Dementia; Non Pharmacological Intervention
Keywords: Non Pharmacological intervention; Alzheimer Disease, Early Onset; Parkinsons Disease with Dementia; Music Therapy
MeSH Terms: conditions — Alzheimer Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Multicenter observational pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- patient with early-onset Alzheimer's disease (AD) (Experimental): patients followed up at the Centre Mémoire de Ressources et de Recherche (CMRR) of Montpellier, over 60 with Alzheimer's disease who have cognitive impairment based on an MMSE (Mini Mental State Examination) ≥ 20 and live at home with a relative
  Interventions: Behavioral: neuropsychologist interview; Behavioral: questionnaire
- patients with parkinson's disease (PD) (Active Comparator): patients followed up at the Center Expert Parkinson of Montpellier (CEPMo), over 60 with Parkinson's disease who have cognitive impairment based on an MMSE (Mini Mental State Examination) ≥ 20 and live at home with a relative
  Interventions: Behavioral: neuropsychologist interview; Behavioral: questionnaire
- Healthy control (Active Comparator): Subjects aged over 60, with no known neurodegenerative disease, living at home with a relative in the Hérault département.
  Interventions: Behavioral: neuropsychologist interview; Behavioral: questionnaire

INTERVENTIONS:
Behavioral: neuropsychologist interview — It will take place either at the hospital or at the participant's home.
  This interview will consist of :
  * socio-demographic data collection
  * neuropsychological tests:
    * MMSE test (Mini Mental State Examination) cognitive function
    * RL-RI-16 test (16-item free recall/indexed recall test)
    * BECS test (Semantic knowledge assessment battery )
    * WCST test (Wisconsin Card Sorting Test )
    * Musical Cognition Test
    * Help from the participant's relative to answer certain questions, in particular the MuseEQ-24 questionnaire
Behavioral: questionnaire — The participant answers questionnaires:
  * Questionnaire MusEQ-24 self reported (Music Engagement Questionnaire)
  * Questionnaire BMRQ (Barcelona Reward Music Questionnaire)
  * Questionnaire SHAPS (Snaith-Hamilton Pleasure Scale)
  * Questionnaire LARS (Lille's Apathy Rating Scale)
  * Questionnaire PHQ-9 (Patient Health Questionnaire 9 items)

SUMMARY:
The goal of this Multicenter observational pilot study is to Compare the specifics of musical engagement (behaviors related to music in everyday life) in subjects aged over 60 with Alzheimer s disease, Parkinson s disease and control subjects.

The main questions it aims to answer are:

1. The description of different profiles of musical engagement in early-stage AD, in PD and in healthy elderly subjects.
2. The extent of executive, mnestic and hedonic dysfunctions will impact differently on emotional engagement, autobiographical evocation and sensitivity to musical reward, and will therefore enable distinct profiles to be drawn up.

Participants will have an intervention consisting of an interview with a neuropsychologist lasting approximately 2 hours, including :

* A semi-structured interview to check the participants eligibility and gather demographic data.
* Neuropsychological tests and questionnaires will then be administered.
* A relative of the study participant will help complete questionnaires.

DETAILED DESCRIPTION:
Music therapy appears to be highly relevant as a Non-Medication Intervention in Alzheimer s (AD) and Parkinson s disease (PD). It is said to reduce depressive symptoms following music therapy sessions in dementia . With regard to Parkinson s disease, music therapy brings benefits in terms of motor skills, communication, breathing and emotional aspects. Reviews point to the need to differentiate beneficial effects according to different pathologies.

To date, no study has investigated the evolution of sensitivity to musical reward in AD. Furthermore, no study has discriminated the evolution of musical engagement in several neurodegenerative pathologies.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* 60 years and older
* French-speaking and volunteering for the study
* Living at home with a relative

Alzheimer's disease inclusion criteria:

* Biological diagnosis of probable Alzheimer's disease according to NINCDS-ADRDA criteria (McKhann et al., 1984)
* MMSE greater than or equal to 20

Inclusion criteria Parkinson's disease :

* Diagnosis of Idiopathic Parkinson's disease
* MMSE greater than or equal to 20

Exclusion Criteria:

* No known neurological pathologies (epilepsy and other non-degenerative CNS diseases) or psychiatric disorders (chronic psychosis and psychotic episodes)
* Autistic disorders
* History of stroke or head trauma
* Unstable medical condition (cancer)
* Subject unable to read and/or write
* Hearing impairment without hearing aids
* Refusal of consent after information
* Persons unable to give consent, research carried out in emergency situations, etc.)
* Non-affiliation with a social security scheme
* Person deprived of liberty (by judicial or administrative decision, or forced hospitalization)
* Person under legal protection (guardianship, curatorship, legal protection)
* Person participating in another research project with an exclusion period still in progress

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the specificities of musical engagement (i.e., music-related behaviors in daily life) in Alzheimer's disease, Parkinson's disease, and among a population of healthy old adults. | Baseline
  Global score of informant version of the Music engagement Questionnaire (MusEQ-24) a 24 items questionnaire that delivers an overall score (ranging from 0 to 120) as well as a score for each of its 6 dimensions (ranging from 0 to 5) of musical engagement: Emotion, Daily life, Social, Response, Preferences and Identity. The higher the score, the greater the level of musical engagement.

SECONDARY OUTCOMES:
The comparison of self- and hetero-questionnaires will be carried out within each group for each MUseQ24 dimension | Baseline
  Compare the results of the self-reported and hetero-reported versions of the Musical Engagement Questionnaire.
  Global score of informant version of the Music engagement Questionnaire (MusEQ-24) a 24 items questionnaire that delivers an overall score (ranging from 0 to 120) as well as a score for each of its 6 dimensions (ranging from 0 to 5) of musical engagement: Emotion, Daily life, Social, Response, Preferences and Identity. The higher the score, the greater the level of musical engagement.
Comparison of global cognition between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  Mini Mental State Examination (MMSE) scoring from 0 (minimum) to 30 (maximum), with higher scores indicating better semantic memory function.
Comparison of Executive Function between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  Wisconsin Card Sorting Test (WCST) which assesses executive functioning globally with a rule deduction task. (Scoring from 0 to 6 for the number of correct categories and 0 to 48 for the number of mistakes). The higher the number of categories, the higher the executive functioning. The higher the number of errors, the lower the executive functioning.
Comparison of Episodic Memory Function between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  Free and Cued Recall Test (RL/RI-16), a 16 items tests scoring from 0 (minimum) to 48 (maximum), with higher scores indicating better memory recall.
Comparison of Semantic Memory Function between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  Recognition subtest of the Battery for the Assessment of Semantic Knowledge (BECS) scoring from 0 to 40.
  Higher scores indicate stronger semantic memory abilities, with lower scores reflecting potential deficits in semantic knowledge.
Comparison of Musical Cognition between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  Test of Orientation in Music Therapy (TOM), scoring from 0 to 34 Higher scores represent better musical cognition abilities, while lower scores may indicate reduced cognitive processing of musical information.
Comparison of Semantic Musical Memory between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  The extension of the Test of Orientation in Music Therapy (TOM), scoring from 24 to 120.
  Higher scores represent better musical cognition abilities, while lower scores may indicate reduced cognitive processing of musical information.
Comparison of Sensitivity to musical reward between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  Barcelona Reward Music Questionnaire BRMQ, (scoring 20 to 100, the lower the score the lower the sensitivity to musical reward). It contains 20 items scored on a 5-point Likert scale. It contains 5 dimensions: musical search, emotional evocation, mood regulation, social reward and sensorimotor.
Comparison of Self-assessed musical engagement between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  MusEQ-24, self-reported Global score of informant version of the Music engagement Questionnaire (MusEQ-24) a 24 items questionnaire that delivers an overall score (ranging from 0 to 120) as well as a score for each of its 6 dimensions (ranging from 0 to 5) of musical engagement: Emotion, Daily life, Social, Response, Preferences and Identity. The higher the score, the greater the level of musical engagement.
Comparison of Memory recall during music listening reward between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  MusEQ-24 item 22, hetero-reported (scoring 0 to 5, the lower the score the lower memory recall)
Comparison of emotional experience during music listening during music listening reward between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  MusEQ-24 Emotion subscale, hetero-reported (scoring 0 to 5, the lower the score the lower the emotional experience)
Comparison of Hedonic function reward between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  Snaith-Hamilton Pleasure Scale (SHAPS), a 14 items scale, Score Range: 0 (minimum) to 14 (maximum).
  Higher scores suggest anhedonia, with lower scores indicating a greater capacity for experiencing pleasure.
Comparison of Affective blunting between Alzheimer's, Parkinson's and healthy elderly groups | Baseline
  Emotional intensity subscale of Lille's Apathy Rating Scale (LARS) a 33 items scale. The LARS is divided into 9 subscales, each scoring -4 to +4.
  Higher scores reflect greater affective blunting (reduced emotional intensity), while lower scores suggest a more typical range of emotional responses.
Comparison of Depression symptoms | Baseline
  Patient Health Questionnaire 9 items (PHQ-9). Score Range: 0 (minimum) to 27 (maximum), each item is rated from 0 to 3 Score Interpretation: Higher scores indicate more severe depressive symptoms, with lower scores suggesting fewer depressive symptoms or none at all.
Correlation between the Barcelona Reward Music Questionnaire (BMRQ) and the Wisconsin Card Sorting Test (WCST) for each group | Baseline
  correlation coefficient R
Correlation between the Barcelona Reward Music Questionnaire (BMRQ) and the 16-item free recall/indexed recall test (RL/RI- 16) for each group | Baseline
  correlation coefficient R
Correlation between Barcelona Reward Music Questionnaire (BMRQ) and Lille's Apathy Rating Scale (LARS) subscale for each group | Baseline
  correlation coefficient R
Correlation between the Barcelona Reward Music Questionnaire (BMRQ) and the Snaith-Hamilton Pleasure Scale (SHAPS) for each group | Baseline
  correlation coefficient R
Correlation between the Emotion Subscale of the MusEQ 24 hetero-reported version and the Wisconsin Card Sorting Test (WCST) for each group | Baseline
  correlation coefficient R
Correlation between the Emotion subscale of the MusEQ 24 hetero-reported version and the 16-item free recall/indexed recall test (RL/RI- 16) for each group. | Baseline
  correlation coefficient R
Correlation between the Emotion subscale of the MusEQ 24 hetero-reported version and the Lille's Apathy Rating Scale (LARS) subscale for each group | Baseline
  correlation coefficient R
Correlation between the Emotion Subscale of the MusEQ 24 hetero-reported version and the Snaith-Hamilton Pleasure Scale (SHAPS) for each group | Baseline
  correlation coefficient R
Correlation between Item 22 of the MusEQ-24 hetero-reported version and Wisconsin Card Sorting Test (WCST) for each group | Baseline
  correlation coefficient R
Correlation between item 22 of the MusEQ-24 hetero-reported version with 16-item free recall/indexed recall test (RL/RI- 16) for each group | Baseline
  correlation coefficient R
Correlation between Item 22 of the MusEQ-24 hetero-reported version and the Lille's Apathy Rating Scale (LARS) subscale for each group | Baseline
  correlation coefficient R
Correlation between Item 22 of the MusEQ-24 hetero-reported version and the Snaith-Hamilton Pleasure Scale (SHAPS) for each group | Baseline
  correlation coefficient R

CONTACTS AND LOCATIONS:
Overall Officials: KARIM BENNYS, MD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- France (3):
  - Montpellier Seniors' Association, Montpellier, Hérault
  - CHU de Montpellier - CEPMo, Montpellier, Hérault
  - CHU de Montpellier - CMRR, Montpellier, Hérault

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bian X, Wang Y, Zhao X, Zhang Z, Ding C. Does music therapy affect the global cognitive function of patients with dementia? A meta-analysis. NeuroRehabilitation. 2021;48(4):553-562. doi: 10.3233/NRE-210018. PMID 33967069
- [Background] Zhang Y, Cai J, An L, Hui F, Ren T, Ma H, Zhao Q. Does music therapy enhance behavioral and cognitive function in elderly dementia patients? A systematic review and meta-analysis. Ageing Res Rev. 2017 May;35:1-11. doi: 10.1016/j.arr.2016.12.003. Epub 2016 Dec 23. PMID 28025173
- [Background] van der Steen JT, van Soest-Poortvliet MC, van der Wouden JC, Bruinsma MS, Scholten RJ, Vink AC. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2017 May 2;5(5):CD003477. doi: 10.1002/14651858.CD003477.pub3. PMID 28462986
- [Background] Platel H, Eustache ML, Coppalle R, Viard A, Eustache F, Groussard M, Desgranges B. Boosting Autobiographical Memory and the Sense of Identity of Alzheimer Patients Through Repeated Reminiscence Workshops? Front Psychol. 2021 Feb 15;12:636028. doi: 10.3389/fpsyg.2021.636028. eCollection 2021. PMID 33679562
- [Background] Morris IB, Vasudevan E, Schedel M, Weymouth D, Loomis J, Pinkhasov T, Muratori LM. Music to One's Ears: Familiarity and Music Engagement in People With Parkinson's Disease. Front Neurosci. 2019 Jun 25;13:661. doi: 10.3389/fnins.2019.00661. eCollection 2019. PMID 31293379
- [Background] Machado Sotomayor MJ, Arufe-Giraldez V, Ruiz-Rico G, Navarro-Paton R. Music Therapy and Parkinson's Disease: A Systematic Review from 2015-2020. Int J Environ Res Public Health. 2021 Nov 4;18(21):11618. doi: 10.3390/ijerph182111618. PMID 34770129
- [Background] Loas G, Duru C, Godefroy O, Krystkowiak P. Hedonic deficits in Parkinson's disease: is consummatory anhedonia specific? Front Neurol. 2014 Mar 10;5:24. doi: 10.3389/fneur.2014.00024. eCollection 2014. PMID 24653714
- [Background] Groussard M, Chan TG, Coppalle R, Platel H. Preservation of Musical Memory Throughout the Progression of Alzheimer's Disease? Toward a Reconciliation of Theoretical, Clinical, and Neuroimaging Evidence. J Alzheimers Dis. 2019;68(3):857-883. doi: 10.3233/JAD-180474. PMID 30883343
- [Background] Belfi AM, Moreno GL, Gugliano M, Neill C. Musical reward across the lifespan. Aging Ment Health. 2022 May;26(5):932-939. doi: 10.1080/13607863.2021.1871881. Epub 2021 Jan 14. PMID 33442987